CLINICAL TRIAL: NCT06813092
Title: Effects of a Single Bout of High Intensity, High Velocity Resistance Exercise Compared to Whole-body Electromyostimulation on Cardiometabolic Risk Factors and Markers of Bone Formation and -Resorption in Young Female Dentists.
Brief Title: Effects of Resistance Exercise Compared to Whole-body Electromyostimulation in Young Female Dentists.
Acronym: FeDeBoMa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: FeDeBoMa02; UKER (Other: University Hospital Erlangen, Germany)
Record Dates: First submitted 2025-02-03; First posted 2025-02-06 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-06

CONDITIONS: Osteopenia; Cardiometabolic Conditions
Keywords: biomarkers; bone metabolism; exercise; whole-body electromyostimulation; female dentists
MeSH Terms: conditions — Bone Diseases, Metabolic; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Randomized two-arm cross-over design
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor were not aware of the group status and were not allowed to ask correspondingly
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole-Body Electromyostimulation (Experimental): One single bout of whole-body electromyostimulation (20 min, bipolar, 85 Hz, 350 µs, rectangular, 6s of impulse, 4s of rest)
  Interventions: Other: Whole-Body Electromyostimulation
- Resistance exercise (Active Comparator): High intensity, high velocity resistance exercise (30 min, 5-6 exercises, 3 sets at 60-85% 1RM)
  Interventions: Other: Resistance exercise

INTERVENTIONS:
Other: Whole-Body Electromyostimulation — 20 min of WB-EMS (bipolar, 85 Hz, 350 µs, 6s impulse - 4s impulse break)
  Arms: Whole-Body Electromyostimulation
Other: Resistance exercise — High-intensity/high velocity multiple set resistance exercise
  Arms: Resistance exercise

SUMMARY:
Due to their high workload and unfavorable working position, young female dentists are particularly at risk of cardiometabolic diseases and an early reduction in bone mineral density (BMD). With focus on the latter issue, short bouts of resistance exercise with high strain magnitude and velocity are commonly considered to be a feasible option to prevent bone loss in the early years of young adulthood. In parallel, whole-body electromyostimulation (WB-EMS) a trainings technology able address all main muscle groups simultaneously, however with dedicated exercise intensity might be a time-effective, joint friendly and safe option to maintain BMD in people unable or unmotivated to exercise conventionally. In the present study, we aim to compare the effects of a single session of WB-EMS versus high intensity, high velocity resistance exercise on biomarkers of bone formation (Procollagen type 1 N propeptide, P1NP) and resorption (C-terminal telopeptide of type I collagen, CTX-I). We hypothesize that no clinically relevant different effects on P1NP and CTX-I were determined.

ELIGIBILITY:
Inclusion Criteria:

* female dental students (>3rd semester) or licensed dentists
* no competitive sports background for >2 years
* normal body mass (BMI>18,5 and <25 kg/m2)

Exclusion Criteria:

* more than one resistance exercise session per week (last 12 month)
* whole-body electromyostimulation during the last 12 month
* amenorrhea, oligomenorrhea

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female dentistry students and young dentists
Enrollment: 16 (Actual)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Changes for C-terminal telopeptide of type I collagen from pre- to 15 min post-exercise | Immediately pre-exercise to 15 min post exercise of a single exercise session
  Changes for C-terminal telopeptide of type I collagen (CTX-I) serum levels from pre- to 15 min post-exercise as determined by blood samples

SECONDARY OUTCOMES:
Changes for Procollagen type 1 N propeptide from pre- to 15 min post-exercise | Immediately pre-exercise to 15 min post exercise of a single exercise session
  Changes for Procollagen type 1 N propeptide (P1NP) serum levels from pre- to 15 min post-exercise as determined by blood samples
Changes for resting glucose from pre- to 15 min post-exercise | Immediately pr to 15 min post-exercise of a single exercise session
  Changes for resting glucose serum levels from pre- to 15 min post-exercise as determined by blood samples
Changes for hemoglobin A1c from pre- to 15 min post-exercise | Immediately pre- to 15 min post-exercise of a single exercise session
  Changes for hemoglobin A1c (HBA1C) serum levels from pre- to 15 min post-exercise as determined by blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Kemmler, PhD, Principal Investigator — University Hospital Erlangen, Germany
Locations (2):
- Germany (2):
  - Institute of Radiology, Erlangen
  - Institute of Radiology, University Hospital NErlangen, Erlangen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kemmler W, Bebenek M, von Stengel S, Bauer J. Peak-bone-mass development in young adults: effects of study program related levels of occupational and leisure time physical activity and exercise. A prospective 5-year study. Osteoporos Int. 2015 Feb;26(2):653-62. doi: 10.1007/s00198-014-2918-8. Epub 2014 Oct 7. PMID 25288444